CLINICAL TRIAL: NCT00561223
Title: The Effect of Iloprost on Gas Exchange and Pulmonary Mechanics in Patients With COPD
Brief Title: Iloprost in Gas Exchange/Pulm Mechanics in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: Iloprost
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1024
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension
Keywords: chronic obstructive pulmonary disease; pulmonary hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): This study will examine the hypothesis that iloprost maintains and improves ventilation perfusion matching in patients with COPD as reflected by 1) a constant or reduced alveolar to arterial O2 difference as calculated from the measured arterial blood gases obtained before and after iloprost administration, 2) an improvement in the lung diffusing capacity for carbon monoxide that occurs in the absence of a change in spirometry, 3) an improvement in the ventilatory equivalent for oxygen and CO2 measured by expired gas analysis.
  It is anticipated that a positive result in this pilot study would lead to a larger long-term study examining the effect of iloprost on gas exchange, exercise tolerance and quality of life in patients with COPD.
  Interventions: Drug: iloprost Inhalation; Drug: iloprost

INTERVENTIONS:
Drug: iloprost Inhalation — inhale 2.5 mg, repeat times one
  Other Names: Ventavis
Drug: iloprost — inhaled 2.5 mg, repeat times one
  Other Names: Ventavis

SUMMARY:
The investigators believe that iloprost will improve gas exchange in COPD patients with pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary hypertension and right heart failure can complicate the management of the patient with advanced COPD. Attempts to treat this pulmonary hypertension with systemic vasodilators frequently result in a worsening of ventilation perfusion matching and an increase sense of dyspnea. This study will look at the effect of an FDA approved pulmonary vasodilator, iloprost, on gas exchange and pulmonary mechanics in patients with COPD. Ten clinically stable patients will be enrolled. They will report to the lab on the morning of the study and after an arterial line is placed, pulmonary function measurements and arterial blood gases will be obtained. Iloprost (2.5 mcg via nebulizer) will be administered and the effect upon arterial blood pressure, respiration and arterial saturation will be monitored. Pulmonary function tests (PFTs) and blood gases will be repeated after 30 minutes. Patients who remain clinically stable without evidence of a fall in arterial PO2 or systemic blood pressure would inhale a second dose of 2.5 mcg of iloprost. The patient will be monitored for a minimum of 2 hours after their last dose of iloprost. Primary outcome variable will be the alveolar arterial O2 difference while secondary outcomes will include PAO2, venous admixture, FVC and FEV1, DLCO and ventilatory equivalents for O2 and CO2. All comparisons will be made using Student's t-test with a Bonferroni correction. The number of study patients was chosen on the basis of a power analysis to provide an alpha of 0.05 at a level of 0.9.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 < 65% of predicted and FEV1 to FVC ratio < 70%
* Baseline PAO2 while stable between 60-75 mmHg and
* The ability to provide informed consent

Exclusion Criteria:

* Clinical instability as evidenced by an acute exacerbation requiring an intensification of therapy and/or the need for hospitalization with the preceding 3 months.
* Presence of an additional cause of lung disease as suggested by history, clinical or radiographic findings, or pulmonary function tests
* Presence of left ventricular dysfunction and/or left atrial enlargement by echo, ECHO or catheterization
* Heparin allergy
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2012-10-31 (Actual)

PRIMARY OUTCOMES:
The alveolar arterial O2 difference | One day

SECONDARY OUTCOMES:
PaO2, vital capacity, FEV1, DLCO, ventilatory equivalents for O2 and CO2 | One day

CONTACTS AND LOCATIONS:
Overall Officials: Gary T Kinasewitz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States